CLINICAL TRIAL: NCT04541212
Title: Identification and Evaluation of Patients at Risk of Developing Cardiotoxicity After Receiving Chemotherapy for Breast Cancer, Lymphoma or Leukemia
Acronym: CarChem
Status: Active, not recruiting | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: MHICC-2018-003
Record Dates: First submitted 2020-07-30; First posted 2020-09-09 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Lymphoma; Leukemia
MeSH Terms: conditions — Breast Neoplasms; Lymphoma; Leukemia | interventions — Hematologic Tests; Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Prospective
  Interventions: Diagnostic Test: Cardiac Imaging
- Cohort B: Retrospective/Prospective
  Interventions: Diagnostic Test: Cardiac Imaging; Other: Data Collection

INTERVENTIONS:
Diagnostic Test: Cardiac Imaging — Cardiac Imaging: echography, ECG, MRI Blood tests: Lipid profile, hs-CRP, metabolic markers, HDL functionality, pharmacogenetic testing (optional), hematocrit, pregnancy test
  Other Names: Blood tests
Other: Data Collection — Collection of retrospective data
  Groups: Cohort B

SUMMARY:
This is an observational study of the occurrence of cardiac toxicity in patients with breast cancer,lymphoma or leukemia receiving chemotherapy including an anthracycline. Patients will be identified at the oncology clinic and will be included in the study if all eligible criteria are met. The study will involve retrospective and prospective evaluations.

Safety will be assessed through reporting of serious adverse events (SAEs) related to study procedures.

DETAILED DESCRIPTION:
The aim of this study is to identify and evaluate cardiotoxicity in patients with diagnosis of breast cancer, lymphoma or leukemia scheduled to receive anthracycline-based chemotherapy (Cohort A: prospective evaluation); and patients undergoing or having received within the last 5 years anthracycline-based chemotherapy (Cohort B: retrospective and prospective evaluations). Part A and B will be conducted in parallel. This study also has the objectif of identifying biomarkers of cardiotoxicity including inflammatory response proteins and clonal hematopoiesis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at time of CT initiation
* Signed informed consent
* Patients with diagnosis of breast cancer,lymphoma or leukemia (including autografted subjects)
* Planned, ongoing or completed (within last 5 years) chemotherapy with anthracycline
* Left ventricular ejection fraction (LVEF) ≥50% pre-chemotherapy
* The participant is willing to undergo CMR scans and all other required study procedures

Exclusion Criteria:

* Known cardiomyopathy and/or LVEF <50%
* Known heart failure
* History of myocardial infarction (MI)
* Clinically significant cardiac valvular disease
* Clinically significant pericardial effusion
* Allografted subjects
* Contraindications to CMR testing (Cohort A & prospective evaluation for Cohort B):

  * Pacemakers, other metallic implants or severe claustrophobia
  * Weight > 135 kg
  * Patients with a history of previous allergic reaction to gadolinium
  * Patients with history of seizure
  * Renal insufficiency (eGFR of < 45ml/min/1.73m2 using the MDRD equation)
  * Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 225 patients enrolled from oncology clinics. Patients will be screened and identified at the oncology clinics. The prospective cardiac evaluations including New York Heart Association (NYHA) functional classification, transthoracic echocardiography, CMR, standard 12-lead electrocardiogram (ECG), cardiac biomarkers, lipid profile & HDL functionality tests will be performed at the Montreal Heart Institute (MHI).
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Myocardial extracellular volume (ECV) | Change from baseline to 3, 6, 12,and 24 months
  Cohort A
Myocardial extracellular volume (ECV) | Change from baseline to prior study entry, 12 and 24 months post study entry.
  Cohort B

SECONDARY OUTCOMES:
Left ventricular (LV) systolic function (global and regional) | Change from baseline to 3, 6, 12,and 24 months.
  Cohort A
Biomarker of myocardial injury (high-sensitivity troponin (hs-cTn)) | Change from baseline to 3, 6, 12,and 24 months.
  Cohort A
Biomarker of elevated LV fitting pressure (N-Terminal-pro-hormone B-type Natriuretic Peptide (NT-proBNP)) | Change from baseline to 3, 6, 12,and 24 months.
  Cohort A
Biomarker of inflammation (high-sensitivity C-reactive protein (hs-CRP)) | Change from baseline to 3, 6, 12,and 24 months.
  Cohort A
Clonal hematopoiesis associated gene mutations. | Change from baseline to 24 months..
  Cohort A
Telomere length measurement | Change from baseline to 24 months..
  Cohort A
Left ventricular (LV) systolic function (global and regional) | Change from study entry to 12 and 24 months.
  Cohort B
Biomarker of myocardial injury (high-sensitivity troponin (hs-cTn)) | Change from study entry to 12 and 24 months.
  Cohort B
Biomarker of elevated LV fitting pressure (N-Terminal-pro-hormone B-type Natriuretic Peptide (NT-proBNP)) | Change from study entry to 12 and 24 months.
  Cohort B
Biomarker of inflammation (high-sensitivity C-reactive protein (hs-CRP)) | Change from study entry to 12 and 24 months.
  Cohort B
Clonal hematopoiesis associated gene mutations. | Change from baseline to 24 months..
  Cohort B
Telomere length measurement | Change from baseline to 24 months..
  Cohort B

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, MD, Principal Investigator — Montreal Heart Institute
Locations (6):
- Canada (6):
  - Centre Hospitalier de l'université de Montréal (CHUM), Montreal, Quebec
  - CIUSSS Ouest de l'ile de Montreal - St-Mary's Hospital, Montreal, Quebec
  - CIUSSS de l'Est-de-l'Île-de-Montréal - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - CIUSSS du Centre-Ouest de l'Île de Montréal - Jewish General Hospital, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - CISSSS de Lanaudière_Hôpital Pierre LeGardeur (referring site), Terrebonne, Quebec (QC)

IPD SHARING:
Plan to Share IPD: No